CLINICAL TRIAL: NCT02813174
Title: Personality Style and Self Compassion in Postpartum Depression: An Online Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i4Health (Other)
Responsible Party: Principal Investigator, Meagan Stanley, Clinical Psychology PhD Candidate, i4Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-018-H
Record Dates: First submitted 2016-06-15; First posted 2016-06-24 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

ARMS (1):
- Automated online Compassionate Mind Training (Experimental)
  Interventions: Behavioral: Compassionate Mind Training from Compassion-Focused Therapy

INTERVENTIONS:
Behavioral: Compassionate Mind Training from Compassion-Focused Therapy

SUMMARY:
The primary aim of this study is to assess the relationship between personality style, self-compassion and depression during pregnancy, to identify psychological risk factors, particularly personality styles, that may contribute to the onset of PPD. Additionally, the study will provide support for the effectiveness of Internet-based Compassionate-Mind Training (iCMT) as a prevention intervention for Postpartum Depression (PPD) for women in the 2nd and 3rd trimester of pregnancy. The study will also assess differences along personality predictors and depression severity as they relate to intervention outcomes (i.e. depression in postpartum and self-compassion) and engagement. The researchers hypothesize that women both at high and low risk for PPD will receive benefits from the intervention, however, those who endorse more maladaptive personality traits will likely engage and benefit less than those who do not endorse these traits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the second and third trimester

Exclusion Criteria:

* Under 18 years of age
* Males
* Women who are not pregnant
* Pregnant women in the first trimester of pregnancy or over 36 weeks pregnant
* Women who likely meet criteria for a Major Depressive Episode
* Women currently in in-person psychological tx

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Change from baseline depression at 6 and 12-weeks postpartum
Vulnerable Personality Style Questionnaire | At baseline
Self Compassion Scale | Change from baseline self-compassion at two weeks post-baseline, and 6 and 12-weeks postpartum

SECONDARY OUTCOMES:
Mini-markers | At baseline
  Saucier's Mini-markers of the Big Five Personality Traits (extraversion, agreeableness, openness, conscientiousness, neuroticism)
Postpartum Depression Predictors Inventory - Revised | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided